CLINICAL TRIAL: NCT02678260
Title: A Phase-I Study of PDR001 Administered to Japanese Patients With Advanced Malignancies
Brief Title: Phase I Study of PDR001 in Patients With Advanced Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X1101
Record Dates: First submitted 2016-01-21; First posted 2016-02-09 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Advanced Malignancies
Keywords: Advanced malignancies; PDR001; Japanese patients; adults
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental): PDR001 will be administered i.v. every two weeks until a patient experiences unacceptable toxicity, progressive disease as per irRC and/or treatment is discontinued at the discretion of the investigator or the patient. The treatment period will begin on Cycle 1 Day 1. For the purpose of scheduling and evaluations, a treatment cycle will consist of 28 days. During the study, cohorts of patients will be treated with PDR001 until the maximum tolerated dose (MTD) is reached or a lower recommended dose (RD) is established.
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — PDR001 is a high-affinity, ligand-blocking, humanized anti-PD-1 IgG4 antibody that blocks the binding of PD-L1 and PD-L2 to PD-1.

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, Pharmacokinetics (PK), and antitumor activity of PDR001 administered intravenous (i.v.) as a single agent to Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by response evaluation criteria in solid tumors (RECIST) version 1.1, who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists
* ECOG Performance Status ≤ 2

Exclusion Criteria:

* Active autoimmune disease
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Prior PD-1- or PD-L1-directed therapy

Other protocol defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 28 days
  cycle = 28 days

SECONDARY OUTCOMES:
PK parameter: AUC | Cycle 1 Day 1 (C1D1), Cycle 3 Day 1 (C3D1)
  To characterize the PK profile of PDR001; cycle = 28 days
Serum concentration vs. time profiles | C1D1, C3D1
  Serum concentration of PDR001 at the scheduled timepoints up to 336 hours after administration
Presence and/or concentration of anti-PDR001 antibodies | Day 1 on from C1 to C6
  To assess the emergence of anti-PDR001 antibodies following one or more intravenous infusions of PDR001.
Objective response rate (ORR) | up to cycle 11; every 2 cycles (8 weeks), after cycle 12; every 3 cycles (12 weeks)
  cycle = 28 days
Duration of response rate (DOR) | up to cycle 11; every 2 cycles (8 weeks), after cycle 12; every 3 cycles (12 weeks)
  cycle = 28 days
Disease control rate (DCR) | up to cycle 11; every 2 cycles (8 weeks), after cycle 12; every 3 cycles (12 weeks)
  cycle = 28 days
PK parameter: Cmax | Cycle 1 Day 1 (C1D1), Cycle 3 Day 1 (C3D1)
  To characterize the PK profile of PDR001; cycle = 28 days
PK parameter: Tmax | Cycle 1 Day 1 (C1D1), Cycle 3 Day 1 (C3D1)
  To characterize the PK profile of PDR001; cycle = 28 days
PK parameter: half-life | Cycle 1 Day 1 (C1D1), Cycle 3 Day 1 (C3D1)
  To characterize the PK profile of PDR001; cycle = 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Kobe, Hyōgo

IPD SHARING:
Plan to Share IPD: No